CLINICAL TRIAL: NCT01833598
Title: The Efficacy of Ultrasound Guided Percutaneous Needle Tenotomy (PNT) Versus Platelet Rich Plasma (PRP) With PNT in the Treatment of Chronic Tendinosis
Brief Title: Percutaneous Needle Tenotomy (PNT) Versus Platelet Rich Plasma (PRP) With PNT in the Treatment of Chronic Tendinosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-189; HSS 2015-189
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Chronic Tendinopathy
Keywords: Chronic tendinopathy; platelet rich plasma; tendonitis; percutaneous tendon tenotomy; pain; shoulder; knee; ankle; foot
MeSH Terms: conditions — Tendinopathy; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNT + PRP (Active Comparator): percutaneous needle tenotomy with peritendinous platelet-rich plasma injection
  Interventions: Procedure: PNT + PRP
- PNT alone (Active Comparator): percutaneous needle tenotomy alone
  Interventions: Procedure: PNT alone

INTERVENTIONS:
Procedure: PNT + PRP — The PNT + PRP group will undergo needle tenotomy under direct and continuous ultrasound guidance with even distribution of PRP into the peritendinous area(s) of PNT around the affected tendon.
  Other Names: percutaneous needle tenotomy with peritendinous platelet-rich plasma injection
  Arms: PNT + PRP
Procedure: PNT alone — The PNT group will undergo needle tenotomy under direct and continuous ultrasound guidance local anesthesia into the affected tendon. 10 minutes after the injection, the ultrasound machine probe will be passed over the areas treated both to evaluate for any structural changes and for any complications.
  Other Names: percutaneous needle tenotomy alone
  Arms: PNT alone

SUMMARY:
Tendinopathy is a clinical syndrome of chronic pain and tendon degeneration that impairs a person's ability to perform daily activities and recreation. Traditional conservative treatments include activity modification, exercises, ice/heat, and medications and corticosteroid injection. A newer treatment is percutaneous needle tenotomy (PNT), in which the affected area is repetitively needled to disrupt pathological tissue and induce bleeding. This turns a nonhealing chronic injury into an acute injury with enhanced healing capability. Another is Platelet Rich Plasma (PRP), whereby patients' own platelets are injected into the affected area, also activating growth factors. There has been promising research in these tendinopathy treatments but more research is needed.

The investigators plan to expand on prior studies to identify a reproducible and efficacious treatment for chronic tendinopathy to reduce pain and improve function and quality of life. Our goal in this study is to assess the efficacy of ultrasound guided (USG) PNT versus PNT with peritendinous PRP as a treatment for chronic tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-100 years
* pain (≥ 5/10 pain on the VAS) that is a direct result of tendinosis as determined by history of injury and study team member physician's best judgment and review of medical records, imaging studies, etc.
* Tendinosis will be confirmed by clinical and ultrasonographic examination by the PI
* ≥3 months of pain after injury that has failed conservative treatments or after corticosteroid (CSI) (must be 3 months after CSI to avoid theoretical tendon rupture)

Exclusion Criteria:

* taking coumadin or other anti-coagulant or anti-platelet medication
* known coagulopathy or bleeding dyscrasia
* current or recent fluoroquinolone prescription
* prior PNT or PRP for the affected tendon(s)
* known systemic illness such as vasculitis, an autoimmune or an inflammatory disease, or uncontrolled diabetes
* presence of other musculoskeletal injury or tendon rupture in the region
* currently are or plan to become pregnant during the study.

  * Patients taking aspirin or NSAIDs are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Improvement in pain based on a visual analog score | Week 2
Improvement in pain based on a visual analog score | Week 4
Improvement in pain based on a visual analog score | Week 6
Improvement in pain based on a visual analog score | Week 8
Improvement in pain based on a visual analog score | Week 12

SECONDARY OUTCOMES:
Activity Level | Week 2
  Function, sleep, general well-being, return to normal activities, work, sports and reduction in pain medication usage.
Activity Level | Week 4
  Function, sleep, general well-being, return to normal activities, work, sports and reduction in pain medication usage.
Activity Level | Week 6
  Function, sleep, general well-being, return to normal activities, work, sports and reduction in pain medication usage.
Activity Level | Week 8
  Function, sleep, general well-being, return to normal activities, work, sports and reduction in pain medication usage.
Activity Level | Week 12
  Function, sleep, general well-being, return to normal activities, work, sports and reduction in pain medication usage.
Complications | Week 2
  bleeding, infection, tendon rupture, allergic reaction, paralysis, or stroke
Complications | Weeks 4
  bleeding, infection, tendon rupture, allergic reaction, paralysis, or stroke
Complications | Weeks 6
  bleeding, infection, tendon rupture, allergic reaction, paralysis, or stroke
Complications | Weeks 8
  bleeding, infection, tendon rupture, allergic reaction, paralysis, or stroke
Complications | Weeks 12
  bleeding, infection, tendon rupture, allergic reaction, paralysis, or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kirschner, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - Department of Rehabilitation Medicine, Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Kaux JF, Forthomme B, Goff CL, Crielaard JM, Croisier JL. Current opinions on tendinopathy. J Sports Sci Med. 2011 Jun 1;10(2):238-53. PMID 24149868
- [Background] Scott A, Ashe MC. Common tendinopathies in the upper and lower extremities. Curr Sports Med Rep. 2006 Sep;5(5):233-41. doi: 10.1097/01.csmr.0000306421.85919.9c. PMID 16934204
- [Background] Fredberg U, Stengaard-Pedersen K. Chronic tendinopathy tissue pathology, pain mechanisms, and etiology with a special focus on inflammation. Scand J Med Sci Sports. 2008 Feb;18(1):3-15. doi: 10.1111/j.1600-0838.2007.00746.x. PMID 18294189
- [Background] Struijs PA, Kerkhoffs GM, Assendelft WJ, Van Dijk CN. Conservative treatment of lateral epicondylitis: brace versus physical therapy or a combination of both-a randomized clinical trial. Am J Sports Med. 2004 Mar;32(2):462-9. doi: 10.1177/0095399703258714. PMID 14977675
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] McShane JM, Shah VN, Nazarian LN. Sonographically guided percutaneous needle tenotomy for treatment of common extensor tendinosis in the elbow: is a corticosteroid necessary? J Ultrasound Med. 2008 Aug;27(8):1137-44. doi: 10.7863/jum.2008.27.8.1137. PMID 18645071
- [Background] McShane JM, Nazarian LN, Harwood MI. Sonographically guided percutaneous needle tenotomy for treatment of common extensor tendinosis in the elbow. J Ultrasound Med. 2006 Oct;25(10):1281-9. doi: 10.7863/jum.2006.25.10.1281. PMID 16998100
- [Background] Housner JA, Jacobson JA, Misko R. Sonographically guided percutaneous needle tenotomy for the treatment of chronic tendinosis. J Ultrasound Med. 2009 Sep;28(9):1187-92. doi: 10.7863/jum.2009.28.9.1187. PMID 19710216
- [Background] Skjong CC, Meininger AK, Ho SS. Tendinopathy treatment: where is the evidence? Clin Sports Med. 2012 Apr;31(2):329-50. doi: 10.1016/j.csm.2011.11.003. PMID 22341021
- [Background] Maffulli N, Longo UG, Denaro V. Novel approaches for the management of tendinopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2604-13. doi: 10.2106/JBJS.I.01744. PMID 21048180
- [Background] Paavola M, Kannus P, Jarvinen TA, Jarvinen TL, Jozsa L, Jarvinen M. Treatment of tendon disorders. Is there a role for corticosteroid injection? Foot Ankle Clin. 2002 Sep;7(3):501-13. doi: 10.1016/s1083-7515(02)00056-6. PMID 12512406
- [Background] Bahr R, Fossan B, Loken S, Engebretsen L. Surgical treatment compared with eccentric training for patellar tendinopathy (Jumper's Knee). A randomized, controlled trial. J Bone Joint Surg Am. 2006 Aug;88(8):1689-98. doi: 10.2106/JBJS.E.01181. PMID 16882889
- [Background] Nguyen RT, Borg-Stein J, McInnis K. Applications of platelet-rich plasma in musculoskeletal and sports medicine: an evidence-based approach. PM R. 2011 Mar;3(3):226-50. doi: 10.1016/j.pmrj.2010.11.007. PMID 21402369
- [Background] Finnoff JT, Fowler SP, Lai JK, Santrach PJ, Willis EA, Sayeed YA, Smith J. Treatment of chronic tendinopathy with ultrasound-guided needle tenotomy and platelet-rich plasma injection. PM R. 2011 Oct;3(10):900-11. doi: 10.1016/j.pmrj.2011.05.015. Epub 2011 Aug 26. PMID 21872551
- [Background] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208
- [Background] de Jonge S, de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. One-year follow-up of platelet-rich plasma treatment in chronic Achilles tendinopathy: a double-blind randomized placebo-controlled trial. Am J Sports Med. 2011 Aug;39(8):1623-9. doi: 10.1177/0363546511404877. Epub 2011 May 21. PMID 21602565
- [Background] Filardo G, Kon E, Della Villa S, Vincentelli F, Fornasari PM, Marcacci M. Use of platelet-rich plasma for the treatment of refractory jumper's knee. Int Orthop. 2010 Aug;34(6):909-15. doi: 10.1007/s00264-009-0845-7. Epub 2009 Jul 31. PMID 19641918
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Naredo E, Cabero F, Beneyto P, Cruz A, Mondejar B, Uson J, Palop MJ, Crespo M. A randomized comparative study of short term response to blind injection versus sonographic-guided injection of local corticosteroids in patients with painful shoulder. J Rheumatol. 2004 Feb;31(2):308-14. PMID 14760802
- [Background] Rutten MJ, Maresch BJ, Jager GJ, de Waal Malefijt MC. Injection of the subacromial-subdeltoid bursa: blind or ultrasound-guided? Acta Orthop. 2007 Apr;78(2):254-7. doi: 10.1080/17453670710013762. PMID 17464615
- [Background] Wolf JM, Ozer K, Scott F, Gordon MJ, Williams AE. Comparison of autologous blood, corticosteroid, and saline injection in the treatment of lateral epicondylitis: a prospective, randomized, controlled multicenter study. J Hand Surg Am. 2011 Aug;36(8):1269-72. doi: 10.1016/j.jhsa.2011.05.014. Epub 2011 Jun 25. PMID 21705157
- [Background] Creaney L, Wallace A, Curtis M, Connell D. Growth factor-based therapies provide additional benefit beyond physical therapy in resistant elbow tendinopathy: a prospective, single-blind, randomised trial of autologous blood injections versus platelet-rich plasma injections. Br J Sports Med. 2011 Sep;45(12):966-71. doi: 10.1136/bjsm.2010.082503. Epub 2011 Mar 15. PMID 21406450
- [Background] Kaux JF, Le Goff C, Seidel L, Peters P, Gothot A, Albert A, Crielaard JM. [Comparative study of five techniques of preparation of platelet-rich plasma]. Pathol Biol (Paris). 2011 Jun;59(3):157-60. doi: 10.1016/j.patbio.2009.04.007. Epub 2009 May 28. French. PMID 19481375
- [Background] Koh ES, Williams AJ, Povlsen B. Upper-limb pain in long-term poliomyelitis. QJM. 2002 Jun;95(6):389-95. doi: 10.1093/qjmed/95.6.389. PMID 12037247
- [Derived] Kirschner JS, Cheng J, Hurwitz N, Santiago K, Lin E, Beatty N, Kingsbury D, Wendel I, Milani C. Ultrasound-guided percutaneous needle tenotomy (PNT) alone versus PNT plus platelet-rich plasma injection for the treatment of chronic tendinosis: A randomized controlled trial. PM R. 2021 Dec;13(12):1340-1349. doi: 10.1002/pmrj.12583. Epub 2021 Apr 28. PMID 33644963